CLINICAL TRIAL: NCT04606121
Title: The Benefit of Enhanced Day Care of Traditional Chinese Medicine: A Retrospective Study of Medical Records
Status: Completed | Type: Observational
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: TCHIRB-10905008-E
Record Dates: First submitted 2020-10-23; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-07

CONDITIONS: Chemotherapy-Induced Change
MeSH Terms: interventions — Massage; Tai Ji

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: enhanced day care of TCM include acupuncture, massage, tai ji quan, TCM herbal medicine — acupuncture twice in enhanced day care of TCM massage twice in enhanced day care of TCM tai ji quan one time in enhanced day care of TCM TCM herbal powder three times a day

SUMMARY:
We collected medical records since June 2017 to November 2019., used pair-T test for questionnaire of CTCAE, BFT-I, WHOQOL to evaluate the benefit of enhanced day care of TCM for cancer patients.

DETAILED DESCRIPTION:
using TCM method as Complementary and Alternative Medicine is worldwide. we collected medical records that using TCM methods for adverse event from cancer therapies. we used CTCAE BFI-T and WHOQOF-BREF to evaluate the benefit.

ELIGIBILITY:
Inclusion Criteria:

- The medical records since June 2017 to December 2019 needed to meet the following criterial: (1)age>20 years old, (2)diagnosis meet ICD10:C00.0-C97 (3) needed to do Taiwan brief version of Common Terminology Criteria for Adverse Events Version4.0(Taiwan brief version scale of CTCAE), scale of the Taiwanese Version of the Brief Fatigue Inventory(BFI-T) and scale of the World Health Organization Quality of Life-BREF(WHOQOL-BREF), and those scales needed to be done pretest when patient came to the clinics and posttest when case end.

Exclusion Criteria:

- The subjects will be excluded if they do not complete pretest and posttest of the following scales:(1) Taiwan brief version scale of CTCAE, (2) BFI-T scale (3) WHOQOL-BREF scale

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cancer patients who needed to accept surgery, or chemotherapy, or radiotherapy, or other conventional cancer therapy
Sampling Method: Non-Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-06-11 (Actual)

PRIMARY OUTCOMES:
scale of Taiwan brief version of Common Terminology Criteria for Adverse Events Version4.0(Taiwan brief version scale of CTCAE) | 2020
  for chemotherapy related adverse effects in Taiwan

SECONDARY OUTCOMES:
scale of the Taiwanese Version of the Brief Fatigue Inventory(BFI-T) | 2020
  evaluate the level of fatique
scale of the World Health Organization Quality of Life-BREF(WHOQOL-BREF) | 2020
  evaluate QOL

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei city hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu HA, Chen CH, Hsieh MH, Wu YC, Chiu JP, Huang CJ, Hsu CH. The Benefit of Enhanced Daycare of Traditional Chinese Medicine for Cancer Treatment Related Adverse Events: A Retrospective Study of Medical Records. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211025634. doi: 10.1177/15347354211025634. PMID 34142595